CLINICAL TRIAL: NCT03951571
Title: Efficacy and Safety of Anlotinib Hydrochloride (AL3818) in Postoperative Adjuvant Therapy for High-grade Soft Tissue Sarcoma -- A Prospective, Randomized, Double-blind, Placebo-controlled, Multicenter Phase II Clinical Trail
Brief Title: Efficacy and Safety of Anlotinib in Adjuvant Therapy for High-grade Soft Tissue Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Chunmeng Wang, Director, Head of Musculoskeletal Oncology, Principal Investigator, Clinical Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB1902197-8
Record Dates: First submitted 2019-05-10; First posted 2019-05-15 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Soft Tissue Sarcoma Adult; High Grade Sarcoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Anlotinib Gruop (Experimental)
  Interventions: Drug: Anlotinib Hydrochloride
- Placebo Group (Placebo Comparator)
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Anlotinib Hydrochloride — Before breakfast, take an Anlotinib hydrochloride placebo once a day, 12 mg (1 pill) at a time. Continuous oral administration for two weeks and stop for one week. Three weeks (21 days) for a treatment cycle. The total treatment cycles is six.
  Arms: Anlotinib Gruop
Drug: Placebo Oral Tablet — Before breakfast, take an placebo once a day, 1 pill at a time. Continuous oral administration for two weeks and stop for one week. Three weeks (21 days) for a treatment cycle. The total treatment cycles is six.
  Arms: Placebo Group

SUMMARY:
To evaluate the efficacy and safety of Anlotinib Hydrochloride Capsule combined with Best Supportive Therapy in the adjuvant treatment of patients with high-grade soft tissue sarcoma after operation, as compared with placebo combined with Best Supportive Therapy.

ELIGIBILITY:
Inclusion Criteria:

* 1.High-grade soft tissue sarcoma patients without standard adjuvant chemotherapy after surgery. Mainly includes: liposarcoma(except for Myxoid/round cell liposarcoma), leiomyosarcoma, malignant peripheral nerve sheath tumor, fibrosarcoma, clear cell sarcoma, alveolar soft part sarcoma, angiosarcoma, epithelioid sarcoma, malignant solitary fibrous tumor and so on. Except for rhabdomyosarcoma, gastrointestinal stromal tumors, dermatofibrosarcoma protuberans, Ewing sarcoma/primary neuroectodermal tumors, inflammatory myofibroblastoma, malignant mesothelioma.

  2.The postoperative microscopic margin was negative and the pathological diagnosis was high-grade soft tissue sarcoma. The diagnosis was completed by pathologists, and the pathological specimens were confirmed by the research center.

  3.The age is ≥18 years old, the ECOG score is ≤2, and the estimated survival time is more than 3 months.

  4.Examinations meet the following criteria:
  1. Blood routine examination: HB ≥ 100g/L(no blood transfusion within 14 days); ANC ≥ 1.5×10^9 /L; PLT ≥ 80×10^9 /L
  2. Other examinations: Cr ≤ upper limit of normal value (ULN); BIL ≤ ULN; ALTAST ≤ 1.5 × ULN (for patients with liver metastasis ≤ 5 × ULN); fasting triglyceride ≤3.0mmol/L; fasting cholesterol ≤7.75mmol/L;
  3. Doppler ultrasound assessment: LVEF ≥ 50%. 5. Females should agree to use contraceptives (such as intrauterine devices (IUD), birth control pills or condoms) during the study period and 6 months after the end of study and the serum or urine pregnancy test was negative within 7 days prior to study enrollment and must be non-lactating; Males should agree to use contraception during the study period and within six months after the end of the study period.

  6.Patients should participate in the study involuntarily, sign the informed consent, and have good compliant and agree to be followed up.

Exclusion Criteria:

* 1. Patients who have received targeted therapy of vascular endothelial growth inhibitors, such as sunitinib, sorafenib, bevacizumab, imatinib, famitinib and apatinib, etc.

  2. Patients who have malignant tumors previously or concomitantly, except for cured skin basal cell carcinoma and cervical carcinoma in situ; 3. Those who participated in other drug clinical trials within 4 weeks; 4. Those who received chemotherapy within 4 weeks. 5. Those who received anticancer therapy previously and have toxic reactions of NCI-CTC AE grade > grade 1 now; 6. Patients who have multiple factors affecting oral medication (such as inability to swallow, Post-gastrointestinal resection, chronic diarrhea and intestinal obstruction, etc.); 7. Patients who have brain metastases, spinal cord compression, cancerous meningitis, or screening CT or MRI findings of brain or pia mater disease.

  8. Patients have any serious or uncontrolled disease, such as:
  1. Unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within 6 months before randomization, severe uncontrolled arrhythmia; patients with unsatisfactory blood pressure control (systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg);
  2. Active or uncontrolled severe infections;
  3. Liver diseases such as cirrhosis, decompensated liver disease and chronic active hepatitis;
  4. Poor control of diabetes mellitus (FBG > 10mmol/L);
  5. Urinary routine examination showed that urinary protein (++) and confirmed by the 24-hour urinary protein quantification(>1.0 g); 9. Long-term unhealed wound or fracture 10. Patients with bleeding tendency (e.g. active gastrointestinal ulcer) or treated with anticoagulants or vitamin K antagonists such as warfarin, heparin or their analogues.

  11. Arterial or venous thrombosis occurred before the first dose, such as cerebrovascular accidents (including transient ischemic attacks), deep vein thrombosis, and pulmonary embolism.

  12. Those who have a history of psychotropic drug abuse and are unable to get rid of or have mental disorders.

  13. Those who have a history of immunodeficiency, including HIV positive or other acquired, congenital immunodeficiency disorders, or organ transplantation.

  14. According to the investigator's assessment, there are serious concomitant diseases that endanger the safety of the patient or affect the patient's completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2019-05-13 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
DFS | 2 years
  Disease Free Survival
1-year and 2-year DFR | 2 years
  1-year and 2-year disease-free survival rates

SECONDARY OUTCOMES:
OS | 2 years
  Overall Survival
LRFS | 2 years
  Local Recurrence Free Survival
DMFS | 2 years
  Distant Metastasis Free Survival

CONTACTS AND LOCATIONS:
Overall Officials: Wangjun Yan, Principal Investigator — Fudan University
Locations (5):
- China (5):
  - Cancer Hospital of Sun Yat-sen, Guangzhou, Guangdong
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - Zhengjiang Cancer Hospital, Hangzhou, Zhejiang
  - Fudan University Shanghai Cancer Center, Shanghai
  - The Six People's Hospital Affiliated to Shanghai Jiao Tong University, Shanghai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang C, Hu X, Yang L, Xu Y, Zheng B, Yang J, Liao Z, Sun Z, Zhang S, Yu L, Yan Y, Chen Y, Fujiwara T, Zhang J, Buhtoiarov IN, Sun Y, Yan W. Anlotinib versus Placebo as Adjuvant Therapy for Localized High-Grade Soft-Tissue Sarcomas: A Phase II, Double-Blinded, Randomized Controlled Trial. Clin Cancer Res. 2025 Apr 1;31(7):1194-1203. doi: 10.1158/1078-0432.CCR-24-2531. PMID 39918552